CLINICAL TRIAL: NCT02839018
Title: Nutrient Pattern Analysis in Critically Ill Patients Using Omics Technology (NAChO): A Prospective Single-center Observational Trial
Brief Title: Nutrient Pattern Analysis in Critically Ill Patients (NAChO)
Acronym: NAChO
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Nestec Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: NAChO
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Intensive Care Unit (ICU) Acquired Weakness (ICU - AW); Muscle Weakness
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, Urine, Muscle biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Central nervous system (CNS) group: n=50 patients with presumed low prevalence of ICU-AW
- Severe sepsis/shock group: n=50 patients with presumed high prevalence of ICU-AW

SUMMARY:
Little is known about nutritional Parameters that potentially influence the course of intensive-care unit acquired weakness (ICU - AW). The investigators aim to elucidate the nutritional profiles in blood, urine and muscle in respective patients at risk.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Written informed consent obtained from the patient's legal representative and later from the patients (as soon as possible)
* Individuals diagnosed with severe head trauma or intracerebral hemorrhage ("central nervous system group") or with severe sepsis/ septic shock ("Sepsis group") at any time from ICU admission until day 5 (i.e. day of screening)
* Patient on the ICU for ≥ 5 days ("ICU long stayer")

Exclusion Criteria:

* Language other than German or French
* Institutionalized Individuals (e.g. prisoners, severe pre-existing mental incapacity)
* Patients with known pre-existing neurological or psychiatric disease that will make informed consent likely impossible
* Patients with known pregnancy or known to be lactating will not be included to the investigation. Due to the observational/ diagnostical nature of the study, a pregnancy test will not be performed.
* Patients on extracorporeal membrane oxygenation (ECMO)
* Clinical signs of pre-existing malnutrition (Body mass index <18)
* Pre-existing evidence for history of anorexia or bulimia
* Parenteral nutrition received within last 5 days (for more than 12 hours) or evidence for parental nutrition needed within next 7 days
* Terminal disease (i.e. life expectancy <14 days)
* Patients with active malignancy
* Patients on biologicals interfering with metabolism (e.g. infliximab)
* Patients on chronic steroid medication (i.e. prednisone equivalent dose >10mg/day)
* Patients on neuromuscular blocking agents on a regular basis (i.e. on a repetitive basis within last 48 hours or evidence for need within next 7 days)
* At screening (day 5): prescribed caloric intake substantially higher (i.e. > 150% of caloric need of indirect calorimetry) than indirect calorimetric results (in intubated patients) or i.e. standard-of-care (25 Kcal/kg body weight/day)
* Severe adipositas defined as BMI >40
* Known pre-existing allergy to standard enteral formulae
* Subject previously enrolled to an interventional trial that is not considered standard-of-care (e.g. investigation of new medication/drug or medical devices)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill patients with severe Sepsis/shock ("Sepsis Group") or intracerebral conditions (CNS Group)
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Differences in blood nutrient levels over time in patients with/without ICU-AW (i.e. "ICU-AW group" vs. "no-ICU-AW group". Primary comparison of interest is between day 14 vs. day 6. | days 6 to 14
Differences in blood nutrient levels over time in patients in "sepsis group" vs. "CNS group". Primary comparison of interest is between day 14 vs. day 6. | days 6 to 14

SECONDARY OUTCOMES:
Differences in urine nutrient levels over time in patients with/ without ICU-AW (i.e. "ICU-AW group" vs. "no-ICU-AW group". Primary comparison of interest is between day 14 vs. day 6. | days 6 to 14
Differences in urine nutrient levels over time in patients in "sepsis group" vs. "CNS group". Primary comparison of interest is between day 14 vs. day 6. | days 6 to 14
Subgroup analysis: differences in nutrient levels at day 14 vs. day 6 in muscle biopsy samples of ICU long stayer patients in study groups (i.e. "ICU-AW" vs. "no-ICU-AW" and "Sepsis" vs. "CNS"). | days 6 to 14

CONTACTS AND LOCATIONS:
Overall Officials: Joerg C Schefold, MD, Principal Investigator — Inselspital, Bern University Hospital; Jukka Takala, MD, Study Chair — Inselspital, Bern University Hospital; Stephan M Jakob, MD, Study Chair — Inselspital, Bern University Hospital
Locations (1):
- Inselspital, Dept of Intensive Care Medicine, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No